CLINICAL TRIAL: NCT01753830
Title: A Multi Center, Randomized, Double Blind, Saline Controlled Study of a Single Injection of Durolane® Versus a Single Injection of Phosphate Buffered Saline (PBS) to Treat Pain Associated With Osteoarthritis of the Knee
Brief Title: Durolane Versus Phosphate Buffered Saline (PBS) in Knee Osteoarthritis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated early due to decision by sponsor
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 35GA1203
Record Dates: First submitted 2012-12-12; First posted 2012-12-20 (Estimated); Results first posted 2020-09-30 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2020-09

CONDITIONS: Knee Osteoarthritis
Keywords: Double-blind; Randomized; Intraarticular injection; Hyaluronic acid; Placebo; Knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Durolane (Experimental): Single intraarticular injection of Durolane
  Interventions: Device: Durolane
- PBS (Placebo Comparator): Single intraarticular injection of PBS
  Interventions: Device: PBS

INTERVENTIONS:
Device: Durolane — 4.5 mL
  Arms: Durolane
Device: PBS — 4.5 mL
  Arms: PBS

SUMMARY:
The purpose of the study is to determine whether a single intra-articular injection of Durolane 4.5 mL is superior to a single injection of PBS 4.5 mL for the relief of joint pain in patients with osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≤ 35 kg/m2
* Symptomatic osteoarthritis (OA) of the knee
* K L severity grade 1 or 2
* If bilateral OA, contralateral knee K L severity grade 0 or 1

Exclusion Criteria:

* Has clinically apparent tense effusion of the index knee
* Has had surgery on the symptomatic knee within the previous 12 months or arthroscopy in the index knee in the past 3 months
* Has any painful orthopedic disorders of the back or hip
* Has a joint disorder other than osteoarthritis in the index knee

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nebojsa Skrepnik, MD, PhD, Principal Investigator — Tucson Orthopaedic Institute
Locations (25):
- United States (25):
  - Anniston, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Hot Springs, Arkansas
  - Beverly Hills, California
  - El Cajon, California
  - Boulder, Colorado
  - Danbury, Connecticut
  - Trumbull, Connecticut
  - Lauderdale Lakes, Florida
  - Pinellas Park, Florida
  - South Miami, Florida
  - Boise, Idaho
  - Meridian, Idaho
  - Evansville, Indiana
  - New Orleans, Louisiana
  - Wheaton, Maryland
  - Kalamazoo, Michigan
  - Springfield, Missouri
  - Oklahoma City, Oklahoma
  - Duncansville, Pennsylvania
  - Wyomissing, Pennsylvania
  - Charleston, South Carolina
  - Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Durolane: Single intraarticular injection of Durolane
  Durolane
- Phosphate Buffered Saline (PBS): Single intraarticular injection of PBS
  PBS
Period: Overall Study
Arm/Group | Durolane | Phosphate Buffered Saline (PBS)
Started | 37 | 38
Completed | 30 | 35
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Durolane | Phosphate Buffered Saline (PBS) | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (8.89) | 59.6 (8.94) | 58.7 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 16 | 19 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 31 | 33 | 64
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 37 | 38 | 75

OUTCOME MEASURES:

1. Primary Outcome: Average Change in WOMAC VAS Pain Score From Week 6 to Week 30
Description: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain score (0-100 mm Visual Analogue Scale (VAS)). Lower score mean less pain.
Time Frame: Up to 30 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Durolane | Phosphate Buffered Saline (PBS)
Number analyzed (Participants) | 37 | 38
units on a scale | -32.3 (19.64) | -26.8 (20.17)

ADVERSE EVENTS:
Arm/Group | Durolane | Phosphate Buffered Saline (PBS)
All-Cause Mortality (participants affected / at risk) | 1/37 | 0/38
Serious Adverse Events (participants affected / at risk) | 2/37 | 1/38
Other Adverse Events (participants affected / at risk) | 15/37 | 13/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durolane (N=37) | Phosphate Buffered Saline (PBS) (N=38)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) — Not related to study product or injection procedure; Resulted in death
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) — Not related to study product or injection procedure
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) — Not related to study product or injection procedure
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Not related to study product or injection procedure
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) — Not related to study product or injection procedure; Pre-treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durolane (N=37) | Phosphate Buffered Saline (PBS) (N=38)
Injection site joint pain (General disorders) | 2 (2) | 0 (0) — Definitely, probably, or possibly related to the study product and/or injection procedure
Injection site pain (General disorders) | 3 (3) | 2 (2) — Definitely, probably, or possibly related to the study product and/or injection procedure
Injection site erythema (General disorders) | 0 (0) | 2 (2) — Definitely, probably, or possibly related to the study product and/or injection procedure
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) — Not related to study product or injection procedure
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) — Not related to study product or injection procedure
Joint effusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) — One event in Durolane group assessed as definitely, probably, or possibly related to the study product and/or injection procedure. The other events not related to study product or injection procedure.
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) — Both events in Durolane group and 1 event in PBS group definitely, probably, or possibly related to the study product and/or injection procedure. 1 event in PBS group not related to study product or injection procedure.
Joint swelling (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3) — 6 events in Durolane group and 1 event in PBS group assessed as definitely, probably, or possibly related to the study product and/or injection procedure. The rest of the events not related to study product or injection procedure.
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) — Not related to study product or injection procedure
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) — 1 event in PBS group assessed as definitely, probably, or possibly related to the study product and/or injection procedure. The rest of the events not related to study product or injection procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes